CLINICAL TRIAL: NCT03978806
Title: Fostering Resilience on Dialysis: A Peer Navigator Study to Improve the Well-being of Latinos on Hemodialysis
Brief Title: Prosperando: Fostering Resilience on Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-0419
Record Dates: First submitted 2019-05-30; First posted 2019-06-07 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Racial/Ethnic Minorities on Dialysis
Keywords: Latino; Hispanic; Dialysis; Navigator; Community health worker
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This will be a pilot RCT (randomized controlled trial) of a 3 month intervention of Latino ESRD patients that will be randomized to one of two arms: 1) PN Arm, in which a bilingual PN provides support with social factors and support with adherence using motivational interviewing during 5 visits or 2) Control (standard care) Arm.
Who Masked: Investigator
Masking Description: The PI will not know arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peer navigator (Active Comparator): The first PN visit will take place within 1-2 weeks of consent. Each of the 5 subsequent PN visits will take place every 1-2 weeks. We expect patients to complete the intervention within 2-3 months of consent. The function of the initial visit is to establish trust and ensure a more personal approach with participants. The community-based PN intervention is grounded in core Latino values (e.g. trust, personalized relationships). The core elements of the PN intervention include patient motivational interviewing as well as patient activation, empowerment (e.g. help with scheduling of healthcare appointments and re-scheduling of missed HD sessions), education (e.g. education of ESKD and need for renal replacement therapy), and social challenges (e.g. access to resources for transportation, benefits, immigration issues). The duration, individuals present during the visit, and content discussed will be documented in the visit form.
  Interventions: Behavioral: Active Comparator: peer navigator
- Control Arm (standard of care) (Placebo Comparator): Standard of care
  Interventions: Other: Placebo Comparator: Control Arm (standard of care)

INTERVENTIONS:
Behavioral: Active Comparator: peer navigator — The intervention is aimed to provide support with social challenges and adherence. The peer navigator will meet with patients to provide support with social challenges and use motivational interviewing to provide support with adherence.
  Arms: peer navigator
Other: Placebo Comparator: Control Arm (standard of care) — Control patients will have met the same inclusion and exclusion criteria as intervention patients.
  Arms: Control Arm (standard of care)

SUMMARY:
Latinos with End-Stage Renal Disease (ESRD) represent 17% of the US adult ESRD community and suffer a disproportionate burden of social challenges that impacts their well-being. With support from the Amos award from the Robert Wood Johnson Foundation (RWJF), the investigators assessed the feasibility of a 1-arm intervention of a 5-visit lay Peer Navigator intervention to support Latino ESRD patients with social challenges and adherence (using motivational interviewing & patient activation). This trial will build on the Amos work as a small Randomized Controlled Trial (RCT). The overall aims of this proposal are to: 1) engage key operational and clinical stakeholders early-on to develop a Peer Navigator-intervention; 2) conduct a pilot RCT of the peer navigator intervention versus standard care to test feasibility and acceptability; and 3) assess the efficacy of the intervention on interdialytic weight gain (primary outcome) as well as health-related quality of life, patient activation, and hemodialysis adherence (secondary outcomes).

DETAILED DESCRIPTION:
The goal of this project is to assess the feasibility and acceptability of a pilot RCT of a culturally tailored peer-navigator (PN) intervention to improve patient-centered and clinical outcomes for Latino patients with end-stage kidney disease (ESKD). We will compare a culturally tailored intervention that includes a PN to control (standard care). In the culturally tailored intervention, the bilingual PN will provide support with social challenges during 5 visits. We will assess the feasibility of (1) referral, (2) recruitment, (3) retention, (4) intervention implementation, and (5) data collection. We will also assess various outcomes including inter-dialytic weight gain and other adherence and patient-centered outcomes.

Specific Aim 1: Conduct a pilot RCT of the peer navigator intervention to assess feasibility, acceptability, as well as outcomes of the proposed peer navigator intervention.

Hypothesis 1: A culturally tailored intervention that consists of a bilingual/culture-concordant peer navigator that provides support with social challenges and support with adherence using motivational interviewing for Latino end-stage kidney disease (ESKD) patients, is feasible and acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Latino
2. Age between 18 and 90 years
3. Diagnosed with end-stage kidney disease
4. Received standard (thrice-weekly HD) for at least 3 months
5. No active substance use (e.g. heavy etoh or opiates)
6. Speak English or Spanish as a primary language
7. Participants must be able to provide informed consent

Exclusion Criteria:

1. Active suicidal intent
2. Present or past psychosis or bipolar disorder
3. Patient to receive kidney transplantation in the next 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Interdialytic weight gain | Data collection 3 months prior to consent (collected retrospectively) and 6 months following study completion
  Inter-dialytic weight gain will be calculated as the monthly average of the difference between the pre-dialysis weight and the weight at the end of the previous dialysis session, divided by determined dry weight, expressed as a percentage of change in weight per day (%Δkg per day).

SECONDARY OUTCOMES:
Kidney Dialysis Quality of Life Short Form - 36 questions | Change from baseline health-related quality of life up to 24 months
  KDQOL(Kidney Disease Quality Of Life) - Short Form 36 (SF-36). The KDQOL Short Form-36 (KDQOL-SF-36), a 36 item survey with five subscales (Physical Component Summary, Mental Component Summary, Burden of Kidney Disease subscale, Symptoms and Problems subscale, and Effects of Kidney Disease on Daily Life). The KDQOL-SF-36 are scored linearly (with higher score indicating better quality of life) on a range of 0-100 using the developer-recommended scoring (available at https://www.rand.org/health-care/surveys_tools/kdqol.html).
Hemodialysis shortening | This will be monitored beginning 3 months prior to enrollment and then 3 months following study completion up to 24 months. Detailed: Monthly for 3 months prior to enrollment, monthly during study and then monthly for 3 months after study completion.
  Hemodialysis shortening: Defined as shortening the hemodialysis session by greater than or equal to 10 minutes.
Hemodialysis adherence | This will be monitored beginning 3 months prior to enrollment and then 3 months following study completion up to 24 months. Detailed: Monthly for 3 months prior to enrollment, monthly during study and then monthly for 3 months after study completion.
  Hemodialysis adherence defined defined as the proportion of monthly scheduled sessions missed (other than for vacation or hospitalization)
Albumin | This will be monitored beginning 3 months prior to enrollment and then 3 months following study completion up to 24 months. Detailed: Monthly for 3 months prior to enrollment, monthly during study and then monthly for 3 months after study completion.
  Albumin
Potassium | This will be monitored beginning 3 months prior to enrollment and then 3 months following study completion up to 24 months. Detailed: Monthly for 3 months prior to enrollment, monthly during study and then monthly for 3 months after study completion.
  Potassium
Phosphorus | Assessed 3 months prior to enrollment, monitored monthly during intervention, and followed for 3 months after intervention
  Phosphorus
Social determinants of health composite survey | Assessed at twice: At time of enrollment and at time of study completion (up to 1 year)
  Several questions from various previously validated surveys that assess social determinants of health.
Self-Efficacy | Assessed at twice: At time of enrollment and at time of study completion (up to 1 year)
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure to assess self-efficacy
Patient Activation Measure | Assessed at twice: At time of enrollment and at time of study completion (up to 1 year)
  Patient Activation Measure has 13 questions, each item is rated on a four-point scale (1 strong disagree to 4 strong agree, with additional 'non-applicable.' Level 1 (less than 47) indicates 'not believing activation is important.' Level 2 (47 to 55.1) indicates 'a lack of knowledge and confidence to take action.' Level 3 (55.2 to 67) indicates 'beginning to take action.' Level 4 (greater than 67) indicates 'taking action.'
Emergency Department visits and hospitalizations | Assessed at twice: At time of enrollment and at time of study completion (up to 1 year)
  Number of Emergency Department (ED) visits and hospitalizations, length of stay
Social Isolation | Assessed twice: At time of enrollment and at time of study completion (up to 1 year)
  PROMIS measure
Qualitative interviews to assess acceptability | Assessed twice: At time of enrollment and at time of study completion (up to 1 year)
  10 participants will be interviewed using semi-structured approach. The results will be a thematic analysis (that ties in the themes and subthemes with illustrative quotes).
Kidney transplantation Questions derived/tailored from two previously published questionnaires. | Assessed twice: At time of enrollment and at time of study completion (up to 1 year)
  Kidney transplantation interest in pursuing, placement on list, receipt of transplantation. Questions were derived and tailored from two studies: Ayanian NEJM 1999;341:1661-9 & Bouleware American J of Transplantation 2005;5:1503-1512. Some are yes/no questions and others are on a Likert Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Fresenius Medical Care Rocky Mountain Dialysis, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share individual participant data at this time. If this changes, this section will be modified.

REFERENCES:
- [Background] Cukor D, Ver Halen N, Asher DR, Coplan JD, Weedon J, Wyka KE, Saggi SJ, Kimmel PL. Psychosocial intervention improves depression, quality of life, and fluid adherence in hemodialysis. J Am Soc Nephrol. 2014 Jan;25(1):196-206. doi: 10.1681/ASN.2012111134. Epub 2013 Oct 10. PMID 24115478
- [Background] Lora CM, Ricardo AC, Brecklin CS, Fischer MJ, Rosman RT, Carmona E, Lopez A, Balaram M, Nessel L, Tao KK, Xie D, Kusek JW, Go AS, Lash JP. Recruitment of Hispanics into an observational study of chronic kidney disease: the Hispanic Chronic Renal Insufficiency Cohort Study experience. Contemp Clin Trials. 2012 Nov;33(6):1238-44. doi: 10.1016/j.cct.2012.07.012. Epub 2012 Jul 27. PMID 22841929
- [Background] Cervantes L, Jones J, Linas S, Fischer S. Qualitative Interviews Exploring Palliative Care Perspectives of Latinos on Dialysis. Clin J Am Soc Nephrol. 2017 May 8;12(5):788-798. doi: 10.2215/CJN.10260916. Epub 2017 Apr 12. PMID 28404600
- [Background] Cervantes L, Linas S, Keniston A, Fischer S. Latinos With Chronic Kidney Failure Treated by Dialysis: Understanding Their Palliative Care Perspectives. Am J Kidney Dis. 2016 Feb;67(2):344-7. doi: 10.1053/j.ajkd.2015.09.026. Epub 2015 Nov 20. No abstract available. PMID 26612276
- [Background] Cervantes L, Chonchol M, Hasnain-Wynia R, Steiner JF, Havranek E, Hull M, Rice J, Kendrick J, Alamillo X, Camacho C, Fischer S. Peer Navigator Intervention for Latinos on Hemodialysis: A Single-Arm Clinical Trial. J Palliat Med. 2019 Jul;22(7):838-843. doi: 10.1089/jpm.2018.0439. Epub 2019 Jan 31. PMID 30702365
- [Background] Cervantes L, Hull M, Keniston A, Chonchol M, Hasnain-Wynia R, Fischer S. Symptom Burden among Latino Patients with End-Stage Renal Disease and Access to Standard or Emergency-Only Hemodialysis. J Palliat Med. 2018 Sep;21(9):1329-1333. doi: 10.1089/jpm.2017.0663. Epub 2018 May 30. PMID 29847204
- [Background] Cervantes L, Zoucha J, Jones J, Fischer S. Experiences and Values of Latinos with End Stage Renal Disease: A Systematic Review of Qualitative Studies. Nephrol Nurs J. 2016 Nov-Dec;43(6):479-493. PMID 30550077
- [Background] Fischer SM, Cervantes L, Fink RM, Kutner JS. Apoyo con Carino: a pilot randomized controlled trial of a patient navigator intervention to improve palliative care outcomes for Latinos with serious illness. J Pain Symptom Manage. 2015 Apr;49(4):657-65. doi: 10.1016/j.jpainsymman.2014.08.011. Epub 2014 Sep 18. PMID 25240788
- [Derived] Cervantes L, Juarez-Colunga E, Powe NR, Flythe JE, Steiner JF, Cukor D, Hasnain-Wynia R, Furgeson S, Golestaneh L, Camacho C, McBeth L, Beaty BL, Shi J, Bacon E, Chonchol M. Community Health Worker Support for Hispanic and Latino Individuals Receiving Hemodialysis: The Navigate-Kidney Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 1;186(1):56-66. doi: 10.1001/jamainternmed.2025.5305. PMID 41203234

DOCUMENTS (1):
  • Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03978806/ICF_000.pdf